CLINICAL TRIAL: NCT04672941
Title: Quality of Life and Preference of COPD Patients After Switching From Tiotropium Monotherapy (Spiriva® Handihaler®) to Dual Therapy With Tiotropium Bromide Plus Olodaterol (Spiolto® Respimat®) Under Real Life Conditions in Greece (ELLACTO II Study)
Brief Title: Quality of Life in Chronic Obstructive Pulmonary Disease (COPD) Patients After Switching to Tiotropium Plus Olodaterol Fixed Dose Combination in Greece
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1237-0098
Record Dates: First submitted 2020-12-14; First posted 2020-12-17 (Actual); Results first posted 2023-11-28 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide; olodaterol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- COPD patients: COPD patients switching from Tiotropium monotherapy to dual therapy with Tiotropium bromide plus Olodaterol.
  All eligible Chronic Obstructive Pulmonary Disease (COPD) patients who had recently switched (within one week) from tiotropium monotherapy (Spiriva® Handihaler®) to dual therapy with tiotropium bromide plus olodaterol (Spiolto® Respimat®), in the Greek private and public sector pulmonary offices and clinics. The follow-up period was 3 months. Participants were visited at baseline (Visit 1) and at 3 months after baseline visit (Visit 2).
  Interventions: Drug: Tiotropium bromide plus Olodaterol

INTERVENTIONS:
Drug: Tiotropium bromide plus Olodaterol — Tiotropium bromide plus Olodaterol
  Other Names: (Spiolto® Respimat®)

SUMMARY:
The primary objective of this non-interventional study (NIS) is to evaluate changes within 3 months in quality of life according to health status evaluated with the COPD Assessment Test (CAT) in COPD patients who have recently switched (within one week) from tiotropium monotherapy (Spiriva® Handihaler®) to dual therapy with tiotropium bromide plus olodaterol (Spiolto® Respimat®), in the Greek private and public sector pulmonary offices and clinics.

ELIGIBILITY:
Inclusion Criteria:

1. Female and male patients ≥40 years of age
2. Patients diagnosed with COPD who have been using tiotropium administered with Spiriva® Handihaler® for at least 3 months before a recent switch (within last week) to a combination therapy with tiotropium bromide plus olodaterol administered with Spiolto® Respimat® has been made
3. Written informed consent prior to participation
4. Patient should be able to read, comprehend and complete study questionnaires

Exclusion Criteria:

1. Patients with contraindications according to Spiolto® Respimat® SmPC
2. Patients who have been treated with inhaled corticosteroids (ICS) as maintenance therapy* or with a Long-acting beta2 adrenoceptor agonist (LABA)/Long-acting muscarinic antagonist (LAMA) combination (free or fixed dose) in the previous 6 weeks

   *Note: patients with temporary corticosteroids (CS) use during acute exacerbations in the previous 6 weeks can enter the study
3. Patients who have been treated with Spiriva® Respimat®, with other LAMA different than Spiriva®, or with a combination of Spiriva®+LABA/ICS in the previous 6 weeks
4. Patients diagnosed with asthma or with asthma COPD overlap syndrome (ACO)
5. Patients for whom availability at the enrolling site during the planned study period of approximately 3 months is not possible
6. Pregnancy and lactation
7. Patients currently listed for lung transplantation
8. Current participation in any clinical trial or any other non-interventional study of a drug or device.

Further exclusion criteria apply.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 1500 patients with chronic obstructive pulmonary disease (COPD) who have recently switched (within one week) from Spiriva® Handihaler® to Spiolto® Respimat® according to the daily clinical practice in the corresponding site, are to be observed.
Sampling Method: Non-Probability Sample
Enrollment: 1396 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2022-02-21 (Actual); Study Completion 2022-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Katsamani, +30 210 8906 108, Study Chair — maria.katsamani.ext@boehringer-ingelheim.com
Locations (2):
- Greece (2):
  - Metropolitan Hospitsal, PNOI Pulmonology Clinic, Athens
  - European Interbalkan Medical Center, Pulmonology Clinic, Thessaloniki

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Also, Researchers can use the following link https://www.mystudywindow.com/msw/datasharing to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
  The data shared are the raw clinical study data sets.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This non-interventional study (NIS) was to evaluate changes within 3 months in quality of life according to health status evaluated with the Chronic Obstructive Pulmonary Disease (COPD) Assessment Test in COPD patients who had recently switched (within one week) from tiotropium monotherapy (Spiriva® Handihaler®) to dual therapy with tiotropium bromide plus olodaterol (Spiolto® Respimat®), in the Greek private and public sector pulmonary offices and clinics.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria.
  Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- COPD Patients: All eligible Chronic Obstructive Pulmonary Disease (COPD) patients who had recently switched (within one week) from tiotropium monotherapy (Spiriva® Handihaler®) to dual therapy with tiotropium bromide plus olodaterol (Spiolto® Respimat®), in the Greek private and public sector pulmonary offices and clinics. The follow-up period was 3 months. Participants visited at baseline (Visit 1) and at 3 months after baseline visit (Visit 2).
Period: Overall Study
Arm/Group | COPD Patients
Started | 1396
Completed | 1388
Not Completed | 8
Not completed — Investigator decision | 1
Not completed — Treatment with Spiolto® Respimat® discontinuation | 2
Not completed — COVID-19 related but no adverse event | 1
Not completed — Adverse Event | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): All patients who were enrolled in the study and have received at least one dose of Spiolto® Respimat®.
Arm/Group | COPD Patients
Number analyzed (Participants) | 1396
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.48 (9.670)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 429
  Male | 967
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Patients' Quality of Life (QoL) According to the Total Score of COPD Assessment Test (CAT) at Month 3
Description: The CAT is a patient-completed questionnaire assessing globally the impact of COPD on health status. It contains 8 items, where each item has a score range from 0 to 5. The CAT score is calculated by summing up the scores from the 8 items. CAT score ranges from 0 to 40. Higher score denotes a more severe impact of COPD on a patient's life. CAT score <10 corresponding to mild impact on patients life is usually considered representing patients without impaired health status.
Time Frame: At baseline and at 3 months after baseline.
Population: Treated Set (TS): All patients who were enrolled in the study and have received at least one dose of Spiolto® Respimat®. Only subjects with both baseline and post baseline values are included.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | COPD Patients
Number analyzed (Participants) | 1342
Score on a scale
  Baseline | 18.41 (6.967)
  Change from baseline | -5.25 (6.281)
Statistical Analysis 1: Comparison: COPD Patients; Test type: Other — Mixed model for repeated measurements (MMRM) assuming random missingness was fitted. The dependent variable was the CAT score at each visit. Visit, Global Initiative for Chronic Obstructive Lung Disease (GOLD) group, smoking habits, pack years, sex, age, and comorbidities appearing at a rate greater than 5% were entered as covariates; Score on a scale = -5.28, 95% CI 2-sided [-5.67 to -4.89] — Least Square Mean for Visit, change from baseline (3 months - baseline) total CAT Score estimates

2. Secondary Outcome: Percentage of Patients With CAT≥10 at Baseline and Month 3
Description: The CAT is a patient-completed questionnaire assessing globally the impact of COPD on health status. It contains 8 items, where each item has a score range from 0 to 5. The CAT score is calculated by summing up the scores from the 8 items. CAT score ranges from 0 to 40. Higher score denotes a more severe impact of COPD on a patient's life. CAT score <10 corresponding to mild impact on patient's life is usually considered representing patients without impaired health status. CAT≥10 refers to impaired health status. The percentages of patients with CAT CAT≥10 at baseline and at Month 3 were reported below.
Time Frame: At baseline and at 3 months after baseline.
Population: Treated Set (TS): All patients who were enrolled in the study and have received at least one dose of Spiolto® Respimat®. The reporting groups below are not mutually exclusive.
Measure: Number; unit: Percentage of participants
Groups:
- COPD Patients - Baseline: All eligible Chronic Obstructive Pulmonary Disease (COPD) patients who had recently switched (within one week) from tiotropium monotherapy (Spiriva® Handihaler®) to dual therapy with tiotropium bromide plus olodaterol (Spiolto® Respimat®), in the Greek private and public sector pulmonary offices and clinics. The follow-up period was 3 months. Participants visited at baseline (Visit 1) and at 3 months after baseline visit (Visit 2).
  Participants with non-missing baseline results were include in this group.
- COPD Patients - Month 3: All eligible Chronic Obstructive Pulmonary Disease (COPD) patients who had recently switched (within one week) from tiotropium monotherapy (Spiriva® Handihaler®) to dual therapy with tiotropium bromide plus olodaterol (Spiolto® Respimat®), in the Greek private and public sector pulmonary offices and clinics. The follow-up period was 3 months. Participants visited at baseline (Visit 1) and at 3 months after baseline visit (Visit 2).
  Participants with non-missing results at 3 months after baseline were include in this group.
Arm/Group | COPD Patients - Baseline | COPD Patients - Month 3
Number analyzed (Participants) | 1396 | 1364
Percentage of participants | 91.76 | 66.12
Statistical Analysis 1: Comparison: COPD Patients - Baseline vs COPD Patients - Month 3; Test type: Other — The logistic generalized estimating equations (GEE) model with CAT response >= 10 as dependent variable. Visit, Chronic Obstructive Lung Disease (GOLD) group, smoking habits, pack years, sex, age, and comorbidities appearing at a rate greater than 5% were entered as covariates and unstructured covariance matrix was used; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 7.186, 95% CI 2-sided [5.745 to 8.987] — Odds ratio for Visit

3. Secondary Outcome: Change From Baseline in the Total European Quality of Life-Visual Analogue Scale (EQ-VAS) at Month 3
Description: The EQ VAS records the patient's self-rated health on a vertical visual analogue scale. EQ-VAS score ranges from 0 to 100 where 0 represents the worst state the patient can imagine and 100 the best. Higher scores indicated better health state.
Time Frame: At baseline and at 3 months after baseline.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | COPD Patients
Number analyzed (Participants) | 1333
Score on a scale | 11.44 (13.225)
Statistical Analysis 1: Comparison: COPD Patients; Test type: Other — Mixed model for repeated measurements (MMRM) assuming random missingness was fitted. The dependent variable was EQ-VAS score. Visit, Global Initiative for Chronic Obstructive Lung Disease (GOLD) group, smoking habits, pack years, sex, age, and comorbidities appearing at a rate greater than 5% were entered as covariates; Score on a scale = 11.80, 95% CI 2-sided [11.00 to 12.60] — Least Square Mean for Visit, mean change from Baseline (3 months - baseline) of EQ-VAS based on non-responder imputation

4. Secondary Outcome: Percentage of Patients With Improved / Worsened Condition Mobility According to the European Quality of Life-5 Dimensions-5 Level (EQ-5D-5L) Questionnaire After 3 Months
Description: EQ-5D-5L descriptive system comprises of 5 dimensions-mobility, self-care, usual activities, pain/discomfort & anxiety/depression. Each dimension has 5 levels: not at all (level 1), mild (level 2), moderate (level 3), severe (level 4), extreme/leading to incapacity (level 5), with highest level corresponding to worst outcome. Subjects had to indicate their health state by choosing the appropriate level from each dimension. The dimension for mobility is reported in this endpoint.
Time Frame: At baseline and at 3 months after baseline.
Population: Treated Set (TS): All patients who were enrolled in the study and have received at least one dose of Spiolto® Respimat®.
Measure: Number; unit: Percentage of participants
Arm/Group | COPD Patients
Number analyzed (Participants) | 1396
Percentage of participants
  Improvement compared to baseline | 44.27
  Deterioration compared to baseline | 2.87
Statistical Analysis 1: Comparison: COPD Patients; Test type: Other — The logistic generalized estimating equations (GEE) model with mobility as dependent variable. Visit, Chronic Obstructive Lung Disease (GOLD) group, smoking habits, pack years, sex, age, and comorbidities appearing at a rate greater than 5% were entered as covariates and unstructured covariance matrix was used; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 4.48, 95% CI 2-sided [3.90 to 5.14] — Odds ratio for Visit (3 months / baseline (reference))

5. Secondary Outcome: Percentage of Patients With Improved / Worsen Condition in Self-care According to the European Quality of Life-5 Dimensions-5 Level (EQ-5D-5L) Questionnaire After 3 Months
Description: EQ-5D-5L descriptive system comprises of 5 dimensions-mobility, self-care, usual activities, pain/discomfort & anxiety/depression. Each dimension has 5 levels: not at all (level 1), mild (level 2), moderate (level 3), severe (level 4), extreme/leading to incapacity (level 5), with highest level corresponding to worst outcome. Subjects had to indicate their health state by choosing the appropriate level from each dimension. The dimension for self-care is reported in this endpoint.
Time Frame: At baseline and at 3 months after baseline.
Population: Treated Set (TS): All patients who were enrolled in the study and have received at least one dose of Spiolto® Respimat®.
Measure: Number; unit: Percentage of participants
Arm/Group | COPD Patients
Number analyzed (Participants) | 1396
Percentage of participants
  Improvement compared to baseline | 30.59
  Deterioration compared to baseline | 3.80
Statistical Analysis 1: Comparison: COPD Patients; Test type: Other — The logistic generalized estimating equations (GEE) model with self-care as dependent variable. Visit, Chronic Obstructive Lung Disease (GOLD) group, smoking habits, pack years, sex, age, and comorbidities appearing at a rate greater than 5% were entered as covariates and unstructured covariance matrix was used; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.64, 95% CI 2-sided [2.35 to 2.96] — Odds ratio for Visit (3 months / baseline (reference))

6. Secondary Outcome: Percentage of Patients With Improved / Worsen Condition Usual Activities According to the European Quality of Life-5 Dimensions-5 Level (EQ-5D-5L) Questionnaire After 3 Months
Description: EQ-5D-5L descriptive system comprises of 5 dimensions-mobility, self-care, usual activities, pain/discomfort & anxiety/depression. Each dimension has 5 levels: not at all (level 1), mild (level 2), moderate (level 3), severe (level 4), extreme/leading to incapacity (level 5), with highest level corresponding to worst outcome. Subjects had to indicate their health state by choosing the appropriate level from each dimension. The dimension for usual activities is reported in this endpoint.
Time Frame: At baseline and at 3 months after baseline.
Population: Treated Set (TS): All patients who were enrolled in the study and have received at least one dose of Spiolto® Respimat®.
Measure: Number; unit: Percentage of participants
Arm/Group | COPD Patients
Number analyzed (Participants) | 1396
Percentage of participants
  Improvement compared to baseline | 43.62
  Deterioration compared to baseline | 4.08
Statistical Analysis 1: Comparison: COPD Patients; Test type: Other — The logistic generalized estimating equations (GEE) model with usual activities as dependent variable. Visit, Chronic Obstructive Lung Disease (GOLD) group, smoking habits, pack years, sex, age, and comorbidities appearing at a rate greater than 5% were entered as covariates and unstructured covariance matrix was used; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 4.46, 95% CI 2-sided [3.89 to 5.12] — Odds ratio for Visit (3 months / baseline (reference))

7. Secondary Outcome: Percentage of Patients With Improved / Worsen Condition Pain/Discomfort According to the European Quality of Life-5 Dimensions-5 Level (EQ-5D-5L) Questionnaire After 3 Months
Description: EQ-5D-5L descriptive system comprises of 5 dimensions-mobility, self-care, usual activities, pain/discomfort & anxiety/depression. Each dimension has 5 levels: not at all (level 1), mild (level 2), moderate (level 3), severe (level 4), extreme/leading to incapacity (level 5), with highest level corresponding to worst outcome. Subjects had to indicate their health state by choosing the appropriate level from each dimension. The dimension for pain/discomfort is reported in this endpoint.
Time Frame: At baseline and at 3 months after baseline.
Population: Treated Set (TS): All patients who were enrolled in the study and have received at least one dose of Spiolto® Respimat®.
Measure: Number; unit: Percentage of participants
Arm/Group | COPD Patients
Number analyzed (Participants) | 1396
Percentage of participants
  Improvement compared to baseline | 43.55
  Deterioration compared to baseline | 4.87
Statistical Analysis 1: Comparison: COPD Patients; Test type: Other — The logistic generalized estimating equations (GEE) model with pain/discomfort as dependent variable. Visit, Chronic Obstructive Lung Disease (GOLD) group, smoking habits, pack years, sex, age, and comorbidities appearing at a rate greater than 5% were entered as covariates and unstructured covariance matrix was used; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.40, 95% CI 2-sided [3.00 to 3.85] — Odds ratio for Visit (3 months / baseline (reference))

8. Secondary Outcome: Percentage of Patients With Improved / Worsen Condition Anxiety/Depression According to the European Quality of Life-5 Dimensions-5 Level (EQ-5D-5L) Questionnaire After 3 Months
Description: EQ-5D-5L descriptive system comprises of 5 dimensions-mobility, self-care, usual activities, pain/discomfort & anxiety/depression. Each dimension has 5 levels: not at all (level 1), mild (level 2), moderate (level 3), severe (level 4), extreme/leading to incapacity (level 5), with highest level corresponding to worst outcome. Subjects had to indicate their health state by choosing the appropriate level from each dimension. The dimension for anxiety/depression is reported in this endpoint.
Time Frame: At baseline and at 3 months after baseline.
Population: Treated Set (TS): All patients who were enrolled in the study and have received at least one dose of Spiolto® Respimat®.
Measure: Number; unit: Percentage of participants
Arm/Group | COPD Patients
Number analyzed (Participants) | 1396
Percentage of participants
  Improvement compared to baseline | 43.27
  Deterioration compared to baseline | 4.01
Statistical Analysis 1: Comparison: COPD Patients; Test type: Other — The logistic generalized estimating equations (GEE) model with anxiety/depression as dependent variable. Visit, Chronic Obstructive Lung Disease (GOLD) group, smoking habits, pack years, sex, age, and comorbidities appearing at a rate greater than 5% were entered as covariates and unstructured covariance matrix was used; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.32, 95% CI 2-sided [2.95 to 3.73] — Odds ratio for Visit (3 months / baseline (reference))

9. Secondary Outcome: Percentage of Patients With Adherence to the Medication
Description: Adherence is measured with the Simplified Medication Adherence Questionnaire (SMAQ), which is a short questionnaire including 6 questions, that assess patient adherence to the medication.
Time Frame: At 3 months after baseline.
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | COPD Patients
Number analyzed (Participants) | 1323
Percentage of participants
  Yes | 67.20
  No | 32.80

10. Secondary Outcome: Total Score in Abbreviated Patient Satisfaction and Preference Questionnaire (PASAPQ)
Description: Calculated from questions 1 to 13 in Part 1 of the PASAPQ. All questions in PASAPQ were answered on a 7-point scale ranging from 1= very dissatisfied to 7 = very satisfied. To calculate the total score, the sum of the 13 items of the two domains (performance and convenience) was transformed to a 0- (least) to 100- (most) point scale which is scaled positively: higher scores represent higher levels of satisfaction.
Time Frame: At 3 months after baseline.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | COPD Patients
Number analyzed (Participants) | 1364
Score on a scale | 78.74 (10.845)

11. Secondary Outcome: Overall Satisfaction of Inhaler
Description: Overall satisfaction according to Question 14 of PASAPQ (Part 1). Question 14 of PASAPQ has a score range from 1= very dissatisfied to 7 = very satisfied.
Time Frame: At 3 months after baseline.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | COPD Patients
Number analyzed (Participants) | 1364
Score on a scale | 6.15 (0.905)

12. Secondary Outcome: Percentage of Patients by Preference for Inhaler
Description: Percentage of patients by preference for inhaler according to Part 2 of the PASAPQ is reported.
Time Frame: At 3 months after baseline.
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | COPD Patients
Number analyzed (Participants) | 1356
Percentage of participants
  Spiriva® Handihaler® | 4.06
  Spiolto® Respimat® | 87.09
  No preference | 8.85

13. Secondary Outcome: Willingness to Continue With Inhaler
Description: According to Part 2 of the PASAPQ; willingness to continue is self-reported by the patient by providing a single value between 1 and 100. 0 indicates that the patient is not willing to continue using the inhaler and 100 indicates that the patient is definitely willing to continue.
Time Frame: At 3 months after baseline.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | COPD Patients
Number analyzed (Participants) | 1356
Score on a scale | 88.39 (14.207)

14. Secondary Outcome: Change From Baseline of Patients' Dyspnea Status According to the Modified Medical Research Council (mMRC) Scale at Month 3
Description: mMRC is a five-level rating scale ranging from 0 to 4 based on the patient's perception of dyspnea in daily activities. A higher score indicates a higher grade of breathlessness.
Time Frame: At baseline and at 3 months after baseline.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | COPD Patients
Number analyzed (Participants) | 1304
Score on a scale | -0.55 (0.776)
Statistical Analysis 1: Comparison: COPD Patients; Test type: Other — Mixed model for repeated measurements (MMRM) assuming random missingness was fitted. The dependent variable was the mMRC score. Visit, Global Initiative for Chronic Obstructive Lung Disease (GOLD) group, smoking habits, pack years, sex, age, and comorbidities appearing at a rate greater than 5% were entered as covariates; Score on a scale = -0.55, 95% CI 2-sided [-0.60 to -0.51] — Least Square Mean for Visit, change from baseline (3 months - baseline) of mMRC based on non-responder imputation

15. Secondary Outcome: Number of Patients Adherence to Medication of COPD Patients According to the Simplified Medication Adherence Questionnaire (SMAQ) Three-months After the Switch
Description: Number of patients adherence to medication of COPD patients according to the Simplified Medication Adherence Questionnaire (SMAQ) three-months after the switch is reported.
Time Frame: At 3 months after baseline.
Population: Treated Set (TS): All patients who were enrolled in the study and have received at least one dose of Spiolto® Respimat®. Only subjects with both baseline and post baseline values and non-missing endpoint values are included.
Measure: Count of Participants; unit: Participants
Arm/Group | COPD Patients
Number analyzed (Participants) | 1356
Participants
  Forget to take the medication for COPD: Yes | 154
  Forget to take the medication for COPD: No | 1162
  Forget to take the medication for COPD: Missing | 40
  Always take your medication for COPD at the indicated time: Yes | 1030
  Always take your medication for COPD at the indicated time: No | 286
  Always take your medication for COPD at the indicated time: Missing | 40
  If feel worse, do you stop taking the medication for COPD?: Yes | 41
  If feel worse, do you stop taking the medication for COPD?: No | 1275
  If feel worse, do you stop taking the medication for COPD?: Missing | 40
  At the last weekend, did you miss your medication?: Yes | 53
  At the last weekend, did you miss your medication?: No | 1263
  At the last weekend, did you miss your medication?: Missing | 40

16. Secondary Outcome: Number of Patients Per Medication Frequency Category According to Simplified Medication Adherence Questionnaire (SMAQ)
Description: Number of patients per medication frequency category according to Simplified Medication Adherence Questionnaire (SMAQ) is reported.
Time Frame: At 3 months after baseline.
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | COPD Patients
Number analyzed (Participants) | 1356
Participants
  Never | 1095
  1-2 times | 201
  3-5 times | 16
  6-10 times | 4
  Missing | 40

17. Secondary Outcome: Days of Missed Medication for COPD
Description: Days of missed medication for COPD is reported.
Time Frame: up to 3 months
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: days
Arm/Group | COPD Patients
Number analyzed (Participants) | 1356
days | 1.55 (4.330)

ADVERSE EVENTS:
Time Frame: From baseline up to 3 months after baseline.
Description: Treated Set (TS): All patients who were enrolled in the study and have received at least one dose of Spiolto® Respimat®.
Arm/Group | COPD Patients
All-Cause Mortality (participants affected / at risk) | 2/1396
Serious Adverse Events (participants affected / at risk) | 2/1396
Other Adverse Events (participants affected / at risk) | 0/1396
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | COPD Patients (N=1396)
Myocardial infarction (Cardiac disorders) | 2
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
COVID-19 (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results.

Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days.

BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-07-09): https://cdn.clinicaltrials.gov/large-docs/41/NCT04672941/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-02): https://cdn.clinicaltrials.gov/large-docs/41/NCT04672941/SAP_001.pdf